CLINICAL TRIAL: NCT02069717
Title: Multi-center, Prospective, Observational Study to Assess the Incidence Rate of the Major Adverse Cardiovascular Events (MACE) and Safety of Fenofibrate (Lipilfen Capsule) Add-on to Statin Therapy in Patients Who Have History of Acute Myocardial Infarction and Are Diagnosed With Metabolic Syndrome
Brief Title: Observational Study to Assess the Incidence Rate of the Major Adverse Cardiovascular Events (MACE) and Safety of Fenofibrate (Lipilfen Capsule)
Status: Withdrawn | Type: Observational
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW_FAMI_001
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months

GROUPS / COHORTS (1):
- Not applicable-observational study: Not applicable-observational study
  Interventions: Other: Not applicable-observational study

INTERVENTIONS:
Other: Not applicable-observational study

SUMMARY:
The purpose of this study was to assess the incidence rate of the major adverse cardiovascular events (MACE) and safety of fenofibrate (Lipilfen capsule) add-on statin therapy in patients who have history of acute myocardial infarction and are diagnosed with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* patients >20 years of age.
* history of acute myocardial infarction
* metabolic syndrome diagnosis

Exclusion Criteria:

* current liver disease or AST or ALT greater than 3 times the upper limit of reference range
* pre-existing gallbladder disease
* moderate to severe renal disorder (serum creatinine >2.5mg/dL)
* pancreatitis diagnosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged more than 20 with history of acute myocardial infarction and diagnosed with metabolic syndrome
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The incidence rate of the major adverse cardiovascular events (MACE) | 24 months
  cardiac death, MI, re-PCI, CABG

SECONDARY OUTCOMES:
The incidence rate of the major adverse cardiac and cerebrovascular event (MACCE) | 24 months
  non-cardiac death, stroke, hospitalization for acute coronary syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- Chonnam national university hospital, Gwangju, South Korea